CLINICAL TRIAL: NCT07199400
Title: Using a Technology Assisted Physical Activity Program to Improve Muscle Strength, Joint Mobility, Standing Time,Self-efficacy and Life Satisfaction of Residents in Institutions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Completed
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202410HM009
Record Dates: First submitted 2025-08-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Mildly Frail; Fragile and More Vulnerable
Keywords: Muscle strength; Joint mobility; Self-efficacy; Life satisfaction; technology assisted physical activity program; residents in institutions; standing time
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using a technology-assisted physical activity program (Experimental): Residents are guided through 26 seated exercises using a digital display and receive real-time feedback. Each set of exercises lasts 30 minutes and is repeated eight times, aiming to improve muscle strength, flexibility, balance, self-efficacy, and life satisfaction.
  Interventions: Behavioral: physical activity program
- Not receiving a technology-assisted physical activity program (No Intervention): Institutional residents can continue their daily physical activities within the facility without digital assistance.

INTERVENTIONS:
Behavioral: physical activity program — Received eight sessions of technology-assisted exercise courses, covering 26 movements in the shoulders, neck, chest, upper limbs and lower limbs, with demonstrations and real-time feedback on movement performance through high-end monitors
  Arms: Using a technology-assisted physical activity program

SUMMARY:
This study aims to examine the effectiveness of a technology-assisted physical activity program on improving muscle strength, joint mobility, standing time, self-efficacy, and life satisfaction among residents in institutions.

With the rapid growth of the aging population in Taiwan and the associated decline in physical function, innovative interventions are urgently needed. The program integrates interactive digital displays to provide safe, guided exercise routines tailored to residents in institutions, with the goal of enhancing both physical and psychological well-being, thereby improving overall quality of life.

DETAILED DESCRIPTION:
Taiwan is rapidly entering a super-aged society, with individuals aged 65 and above projected to exceed 20% of the total population by 2025. Aging is associated with declines in muscle endurance, joint mobility, balance, and functional independence, which severely affect daily living performance. Although aging cannot be prevented, appropriate interventions can slow down functional decline and improve quality of life.

This study used a randomized controlled trial design to investigate the effects of a technology-assisted exercise intervention in long-term care facilities. Residents classified as frail or mildly frail according to the Clinical Frailty Scale were recruited and randomly assigned to either the intervention group (n=26) or the control group (n=25).

The intervention group will participate in eight sessions of a technology-assisted exercise program, consisting of 26 seated movements covering the neck, shoulders, chest, upper and lower limbs. The program, designed by faculty and students from National Taiwan University of Sport, emphasizes safety and accessibility for Residents. Exercises will be demonstrated via an advanced digital display system with real-time feedback, and each session will last approximately 30 minutes. The control group will maintain routine physical activities without digital assistance.

ELIGIBILITY:
Inclusion Criteria:

Suitable for participation in an exercise intervention program. Able to understand and comply with study instructions, willingly participate, and sign an informed consent form.

Exclusion Criteria:

Residents with severe cognitive impairment or unable to cooperate with exercise guidance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Joint Mobility | Baseline and post-intervention (8 weeks).
  Range of motion of upper and lower limb joints measured with goniometer (degrees).
Muscle Strength | Baseline and post-intervention (8 weeks).
  Description: Grip strength measured by dynamometer (kg).
Standing Time | Baseline and post-intervention (8 weeks).
  Description: Maximum duration of standing measured in seconds to assess balance and lower-limb strength.
Self-Efficacy | Baseline and post-intervention (8 weeks).
  Self-efficacy for daily activities assessed using validated self-efficacy scale. Higher scores indicate stronger confidence. scale scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores indicate stronger self-efficacy.
Life Satisfaction | Baseline and post-intervention (8 weeks).
  Global life satisfaction assessed with the Satisfaction with Life Scale (SWLS). Higher scores indicate greater satisfaction. Global life satisfaction assessed with the Satisfaction with Life Scale (SWLS), a 5-item scale scored on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). Higher scores indicate greater life satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University,Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and ethical considerations. Only aggregate results will be reported in publications.